CLINICAL TRIAL: NCT04097405
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, and Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of D-0120 in Healthy Volunteers
Brief Title: Phase I Study of D-0120 to Evaluate Safety and PK/PD Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: IBIO-203
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- D-0120 Dose Ascending Cohorts 1-4 (Active Comparator): D-0120 dose daily for up to 7 days.
  Interventions: Drug: D-0120
- Placebo Dose Ascending Cohorts 1-4 (Placebo Comparator): Placebo dose daily for up to 7 days
  Interventions: Drug: Placebo oral tablet
- D-0120/Uric Acid Lowering Agent Cohort 6 (Experimental): D-0120 in combination with a uric acid lowering agent for up to 7 days of combination therapy
  Interventions: Drug: D-0120

INTERVENTIONS:
Drug: D-0120 — Randomized, Double-Blind, Placebo-Controlled, Multiple Dose and Dose Escalation of D-0120 or Placebo
  Arms: D-0120 Dose Ascending Cohorts 1-4; D-0120/Uric Acid Lowering Agent Cohort 6
Drug: Placebo oral tablet — Randomized, Double-Blind, Placebo-Controlled, Multiple Dose and Dose Escalation of D-0120 or Placebo
  Arms: Placebo Dose Ascending Cohorts 1-4

SUMMARY:
This phase 1 study is a randomized, double-blind, placebo controlled, multiple-dose, dose-escalating study to evaluate the safety, tolerability, PK and PD of D-0120 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be medically documented as healthy at physical examination
* Moderate smokers or non-smokers
* Subjects must be between the ages of 18 and 60
* Subject must have a BMI between 18.0 and 30.0 kg/m2 (inclusive)
* Subjects must have a body weight of 50kg or higher for males and 45kg or higher for females
* Females must be non-pregnant and non-lactating, and either surgically sterile at least 6 months prior to the first study drug administration or post-menopausal for 12 months or greater
* Male subjects who are not vasectomized for at least 6 months, and who are sexually active with non-sterile female partner must be willing to use an acceptable contraceptive method throughout the study and for 90 days after the last study drug administration
* Male subjects with a pregnant partner must agree to use a condom from the first dosing until at least 90 days after the last study administration
* Subjects must have a complete blood count and platelet count within the normal range
* Subjects must have a normal urinalysis
* Subjects must have a normal estimated glomerular filtration rate
* Subjects must have a normal ECG
* Subjects must be able to understand the study procedures, risks involved and be able to comply with the study and follow-up procedures
* Male subjects must be willing not to donate sperm until 90 days following the last study drug administration

Exclusion Criteria:

* Subjects with any history or clinical manifestations of disorders
* Subjects who have any history or suspicion of kidney stones
* Subjects who are HIV, Hep B or Hep C positive
* History of significant allergic reactions to any drug
* Clinically significant ECG abnormalities
* History of significant drug abuse within 1 year prior to screening or use of soft drugs within 3 months prior to screening or hard drugs within 1 year prior to screening
* Subjects who have used prescription dugs, over the counter drugs or herbal remedies within 14 days before day 1
* Positive urine drug screen, alcohol breath at screening
* Subjects had undergone major surgery within 3 months
* Women who are pregnant or breastfeeding
* History of significant alcohol abuse
* Subjects who consumed Seville oranges-or grapefruit-containing food or beverages within 7 days before Day 1 and during the entire study duration.
* Subjects with any condition that, in the judgement of the investigator, would place him/her at undue risk
* Participation in a clinical research study involving the administration of an investigation or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to first dose
* Donation of plasma within 7 days prior to dosing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
The number of subjects with treatment related adverse events as assessed | Reporting of adverse events starts at enrollment through the end of the follow up period (14 days (cohorts 1-4) and 16 days (cohort 6)
  Data will include clinical observations, ECG, clinical chemistry/hematology/urinalysis and vital signs

SECONDARY OUTCOMES:
Time to observed Cmax (Tmax)for D-0120 | Timeframe: Day 1-Day7
  Blood samples will be collected to assess plasma concentrations of D-0120 at a series of timepoints to derive Tmax
Area under the plasma concentration-time curve (AUC) for D-0120 | Day 1-Day 7
  Blood samples will be collected to assess plasma concentration of D-0120 at a series of timepoints to derive AUC
Maximum Observed Plasma Concentration (Cmax) of D-0120 | Day 1-Day 7
  Blood samples will be collect to assess plasma concentrations of D-0120 at a series of timepoints to derive Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No